CLINICAL TRIAL: NCT02398500
Title: An Open-label Single Ascending Dose and Randomized Double-Masked, Ranibizumab Controlled, Safety, Tolerability, and Efficacy Study of Intravitreal LMG324 in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: Safety Tolerability and Efficacy of Intravitreal LMG324 in the Treatment of Neovascular Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Collaborators: Novartis Institutes for BioMedical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LMG324-2201; 2014-005214-37 (EudraCT Number)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: First-in-human; anti-VEGF; neovascular AMD (nvAMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LMG324 (Experimental): SAD: LMG324 administered as a single IVT injection in 1 eye (study eye) in 1 of 4 doses, with 15-day follow-up
  Interventions: Biological: LMG324
- LMG324 + sham (Experimental): Expansion: LMG324 administered as a single IVT injection in 1 eye (study eye), followed by sham injections, until implementation of SoC therapy as specified in the protocol, for 24 weeks
  Interventions: Biological: LMG324; Biological: Sham
- Lucentis + sham (Active Comparator): Expansion: Ranibizumab 0.5 mg administered as monthly IVT injections in 1 eye (study eye) with interim sham injections, for 24 weeks
  Interventions: Biological: Ranibizumab 0.5 mg; Biological: Sham

INTERVENTIONS:
Biological: LMG324 — IVT injection
  Arms: LMG324; LMG324 + sham
Biological: Ranibizumab 0.5 mg — IVT injection
  Other Names: Lucentis®
  Arms: Lucentis + sham
Biological: Sham — Fake injection used for masking purposes
  Arms: LMG324 + sham; Lucentis + sham

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety and tolerability of single ascending doses of LMG324 to determine the maximum tolerated dose (MTD) in neovascular age-related macular degeneration (nvAMD) subjects. Enrollment will be expanded at a safe and tolerated dose in treatment naïve nvAMD subjects to compare a single intravitreal (IVT) dose of LMG324 to ranibizumab 0.5 mg administered every 4 weeks for change from baseline in best-corrected visual acuity (BCVA) at Week 12 (Day 85).

DETAILED DESCRIPTION:
The study will start with a single dose ascending (SAD) phase. LMG324 will be administered on Day 1 with no further treatment until implementation of standard of care (SoC) therapy. SoC therapy is ranibizumab 0.5 mg administered per label. Dose groups will be implemented sequentially to allow for safety review between the current and subsequent dose group. All treatments will be open-label, including ranibizumab used as SoC therapy.

In the enrollment expansion phase, subjects randomized to LMG324 arm will receive a single LMG324 IVT injection on Day 1 followed by sham (fake) IVT injections until implementation of SoC therapy. After implementation, SoC therapy will be applied monthly with sham injections applied at the interim planned visits. The enrollment expansion phase may start at a selected dose level whilst the dose escalation phase is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent, be able to make the required study visits and follow instructions.
* Best corrected visual acuity (BCVA) of 34 letters (approximately 20/200 Snellen or better) in the non-study eye.

SAD population only:

* Subject's study eye must have a choroidal neovascularization (CNV) lesion due to age-related macular degeneration (AMD), either treatment naïve or previously treated, that can be expected to benefit, in the opinion of the investigator, from anti-vascular endothelial growth factor (anti-VEGF) therapy.
* Previously treated eyes must have a history of least 3 administrations of any intravitreal (IVT) anti-VEGF therapeutic for the treatment of CNV with the last injection administered ≥ 1 month prior to the planned administration of the study drug.

Enrollment expansion population only

* Subject's study eye must have untreated and active CNV lesion due to AMD.
* BCVA, between 73 - 23 letters, inclusive (approximate Snellen equivalent 20/40 - 20/320) in the study eye.

Exclusion Criteria:

SAD and enrollment expansion population

* Both eyes: any active ocular or periocular infection or active intraocular inflammation (eg, infectious blepharitis, infectious conjunctivitis, keratitis, scleritis, endophthalmitis).
* Study eye: current vitreous hemorrhage or a history of rhegmatogenous retinal detachment.
* Study eye: uncontrolled glaucoma (intraocular pressure [IOP] >25 mmHg on medication or according to Investigator's judgment).

SAD population only

* Presence of any contraindications, in the Investigator's opinion, to IVT anti-VEGF therapeutic administration.

Enrollment expansion population only

* Study eye: subject has received any approved or investigational treatment for exudative (wet) AMD other than vitamin supplements.
* Study eye: any current or history of macular or retinal disease other than exudative AMD
* Study eye: serous pigment epithelial detachment (PED) under the foveal center or retinal pigment epithelium (RPE) tear/rip.
* Study eye: any concurrent intraocular condition (eg, cataract, diabetic retinopathy) that, in the opinion of the Investigator, could either require medical or surgical intervention during the course of the study.
* Study eye: other ocular diseases that, in the opinion of the Investigator, can compromise the visual acuity
* Study eye: Surgery, as specified in the protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in best corrected visual acuity (BCVA) at Day 85 | Baseline, Day 85

SECONDARY OUTCOMES:
Percentage of LMG324-treated subjects with no identified SoC treatment need up to and including Day 85 | Up to Day 85
Best Corrected Visual Acuity (BCVA) | Up to Day 169
Central subfield thickness total (CSFTtot) | Up to Day 169
Central subfield thickness neuro-retina (CFSTnr) | Up to Day 169
Lesion thickness | Up to Day 169
Subretinal fluid with foveal involvement (SRFfi) thickness | Up to Day 169
Retinal pigment epithelial detachment with foveal involvement (PEDfi) thickness | Up to Day 169
Area of lesion (associated with CNV) | Up to Day 169
Area of CNV within a lesion | Up to Day 169
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | Up to Day 169
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | Up to Day 169
Area under the plasma concentration-time curve from time zero to time 't' where t is a defined time point after administration (AUC0-t) | Up to Day 169
Maximum observed maximum plasma concentration (Cmax) | Up to Day 169
Time to reach the maximum observed plasma concentration (Tmax) | Up to Day 169
Observed maximum plasma concentration following drug administration, by dose (Cmax/D) | Up to Day 169
Area under the plasma concentration-time curve divided by dose (AUC/D) | Up to Day 169
Frequency of subjects with anti-LMG324 antibodies | Up to Day 169

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Scientist I, NIBR, Study Director — Alcon Research
Locations (1):
- Call Alcon Call Center for Trial Locations, Fort Worth, Texas, United States